CLINICAL TRIAL: NCT06735326
Title: A Randomized, Open-Label, Multi-Cohort Study of Fluzoparib Monotherapy or in Combination With Bevacizumab as Neoadjuvant Therapy in Patients With Advanced Ovarian Cancer
Brief Title: Fluzoparib With or Without Bevacizumab for Neoadjuvant Therapy in Advanced Ovarian Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KYLL-202410-008-1
Record Dates: First submitted 2024-11-25; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — fluzoparib; Bevacizumab; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fluzoparib monotherapy (Experimental): Fluzoparib capsules with a treatment cycle of 28 days, for a total of 2 cycles.
  Interventions: Drug: Fluzoparib
- Fluzoparib in combination with Bevacizumab (Experimental): Fluzoparib capsules with a treatment cycle of 28 days, for a total of 2 cycles; in combination with Bevacizumab injection (7.5mg/kg, intravenous infusion, administered once every three weeks), for a total of 2 doses.
  Interventions: Drug: Fluzoparib; Drug: Bevacizumab
- Paclitaxel plus Carboplatin (Active Comparator): Paclitaxel injection plus Carboplatin injection, administered once every three weeks for a total of 3 doses. If there is an allergy to Paclitaxel, it is recommended to replace it with Docetaxel or Liposomal Doxorubicin.
  Interventions: Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Fluzoparib — Fluzoparib capsule (50mg per capsule) 150mg po BID
  Arms: Fluzoparib in combination with Bevacizumab; Fluzoparib monotherapy
Drug: Bevacizumab — Bevacizumab injection (100mg per vial) 7.5mg/kg ivdrip Q3W
  Arms: Fluzoparib in combination with Bevacizumab
Drug: Paclitaxel — Paclitaxel injection 135-175mg/㎡ ivdrip Q3W
  Arms: Paclitaxel plus Carboplatin
Drug: Carboplatin — Carboplatin injection AUC=4-5 ivdrip Q3W
  Arms: Paclitaxel plus Carboplatin

SUMMARY:
This study is a randomized, open-label, multi-cohort, multicenter clinical trial, aimed at evaluating the efficacy and safety of Fluzoparib monotherapy, Fluzoparib in combination with Bevacizumab, and standard chemotherapy (Paclitaxel plus Carboplatin) as neoadjuvant treatments in newly diagnosed, germline BRCA1/2-mutated epithelial ovarian cancer patients (FIGO stage III/IV). The study also aims to assess the efficacy and safety of Fluzoparib as maintenance therapy following surgery and chemotherapy.

The primary endpoint of the study is the objective response rate (ORR) for neoadjuvant therapy, as assessed by the investigator using RECIST v1.1 criteria. Secondary endpoints include R0 resection rate, overall survival (OS), and progression-free survival (PFS). The study will also evaluate the safety, tolerability, and patient-reported outcomes (EQ-5D-5L) across the three treatment cohorts.

ELIGIBILITY:
Inclusion Criteria:

1. The subject voluntarily agrees to participate and signs the informed consent form.
2. Age ≥18 years (calculated as of the date of signing the informed consent).
3. Pathologically diagnosed with newly diagnosed, FIGO stage III-IV high-grade (or moderate/low-grade) serous ovarian cancer, fallopian tube cancer, or primary peritoneal cancer; grade ≥II endometrioid adenocarcinoma of the ovary; Mixed tumors: high-grade serous or ≥II grade endometrioid component must be >50%.
4. The subject has at least one measurable lesion that can be assessed by CT or MRI (RECIST v1.1).
5. According to the investigator's assessment, the patient is unable to achieve R0 resection or cannot tolerate surgery.

   a) Criteria for determining inability to achieve R0 resection include: i. Fagotti laparoscopic score ≥8. ii. If laparoscopic assessment is difficult, an upper abdominal Suidan's CT score ≥3.

   b) Criteria for inability to tolerate surgery include: i. Body mass index (BMI) ≥40. ii. Multiple chronic diseases. iii. Malnutrition or hypoalbuminemia. iv. Moderate to large ascites. v. Newly diagnosed venous thromboembolism. vi. ECOG performance status >2. vii. Other reasons judged by the investigator.
6. Expected survival >12 weeks.
7. ECOG performance status: 0-2.
8. Confirmed germline BRCA1/2 mutations by professional genetic testing.
9. Function of major organs meets the following requirements (no blood products or colony-stimulating factors allowed within 14 days prior to the first dose):

   1. Absolute neutrophil count ≥1.5 × 10^9/L.
   2. Platelet count ≥100 × 10^9/L.
   3. Hemoglobin ≥9 g/dL.
   4. Serum albumin ≥3 g/dL.
   5. Bilirubin ≤1.5 times the upper limit of normal (ULN).
   6. ALT and AST ≤2.5 times ULN, must be ≤5 times ULN in the presence of liver metastases.
   7. Serum creatinine ≤1.5 times ULN, or creatinine clearance ≥60 mL/min (calculated using the Cockcroft-Gault formula).
10. Female patients of childbearing potential must have a negative blood pregnancy test within one week before the first dose and are not breastfeeding. They must agree to use effective contraception during the study and for 6 months after the last dose of Bevacizumab/Fluzoparib/chemotherapy. Pregnancy, if confirmed, must be terminated as soon as possible.
11. The subject is willing to cooperate in completing quality of life surveys during the treatment and follow-up periods and agrees to have the survey results used for clinical research.

Exclusion Criteria:

1. Patients with other untreated malignant tumors within the past 5 years, except for cured skin basal cell carcinoma, cervical carcinoma in situ, and breast cancer without relapse for over 3 years after radical surgery.
2. Patients with untreated central nervous system metastases. Patients who have previously received systemic or curative brain or meningeal metastasis treatment (radiotherapy or surgery) and have stable imaging confirmed for at least 1 month, and have stopped systemic steroid treatment (dosage >10 mg/day prednisone or equivalent) for more than 2 weeks, and have no clinical symptoms, may be included.
3. Patients who have previously received treatment with known or potential PARP inhibitors or Bevacizumab.
4. Patients unable to swallow tablets or with gastrointestinal dysfunction that may affect drug absorption, as judged by the investigator.
5. Patients who have experienced bowel obstruction or gastrointestinal perforation within the last 3 months.
6. Patients with poorly controlled heart conditions or diseases, such as:

   1. NYHA Class II or higher heart failure.
   2. Unstable angina.
   3. Myocardial infarction within 1 year.
   4. Clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention.
   5. QTc >470 ms.
7. Patients with clinically significant bleeding symptoms or a clear bleeding tendency (such as gastrointestinal bleeding, bleeding ulcers, or vasculitis) within 3 months prior to the first dose, or with positive occult blood in the stool at baseline. If positive, it should be rechecked, and if still positive, clinical judgment should be made, including possible gastrointestinal endoscopy if necessary.
8. Patients who have received platelet or red blood cell transfusion within 14 days before starting treatment.
9. Patients with active ulcers, non-healing wounds, or fractures.
10. Patients who have experienced any severe bleeding event graded ≥2 in CTCAE 5.0 within 4 weeks before the first dose.
11. Patients with active infections or unexplained fever >38.5°C during screening or before the first dose.
12. Patients with congenital or acquired immune deficiency (e.g., HIV-infected individuals) or active hepatitis (HBV reference: HBsAg positive, HBV DNA ≥500 IU/ml; HCV reference: HCV antibody positive, HCV RNA > normal upper limit).
13. Patients who have previously received radiotherapy, chemotherapy, hormonal therapy, or molecular targeted therapy, with less than 4 weeks since the last dose of treatment (less than 5 half-lives for oral molecular-targeted agents); patients who have not recovered from treatment-related adverse events (except for hair loss) to ≤1 grade as per CTCAE 5.0.
14. Patients who have experienced arterial thrombosis or ≥grade 3 venous thromboembolic events within 6 months prior to the first dose, such as cerebrovascular accidents (including transient ischemic attacks, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, or pulmonary embolism.
15. Patients with a history of hereditary or acquired bleeding disorders or coagulation dysfunction (e.g., hemophilia, platelet dysfunction, thrombocytopenia, etc.).
16. Patients who may receive other systemic antitumor treatments during the study period.
17. Patients with uncontrolled hypertension, despite antihypertensive treatment (systolic blood pressure ≥150 mmHg or diastolic blood pressure ≥90 mmHg).
18. Pregnant or breastfeeding women, or women planning pregnancy during the study treatment.
19. Patients with other factors, as judged by the investigator, that may lead to the premature termination of the study, such as other severe diseases (including psychiatric disorders) requiring concurrent treatment, severe laboratory abnormalities, or factors related to family or social circumstances that may impact the patient's safety, or the collection of data and samples.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2024-11-27 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | At the end of neoadjuvant treatment. The Fluzoparib monotherapy and Fluzoparib plus Bevacizumab groups will receive 2 cycles of treatment (28 days per cycle). The Paclitaxel plus Carboplatin group will receive 3 cycles of treatment (21 days per cycle).
  The percentage of patients who achieve a complete response (CR) or partial response (PR) as determined by the investigator based on RECIST v1.1 criteria, at the end of neoadjuvant treatment.

SECONDARY OUTCOMES:
R0 resection rate | Immediately after final interval debulking surgery.
  To evaluate the proportion of patients who achieve R0 resection following neoadjuvant therapy.
pCR | Post-surgical pathology (up to 2 weeks post surgery).
  Pathological complete response.
Overall survival (OS) | The time from patient enrollment until the date of death from any cause, assessed up to 120 months.
  The time from patient enrollment to death.
Progression free survival (PFS) | The time from patient enrollment until the date of first documented tumor progression or death from any cause, whichever occurs first, assessed up to 60 months.
  The time from patient enrollment to tumor progression or death.
Safety evaluation | From the start of neoadjuvant therapy to the end of maintenance therapy, assessed up to 30 months.
  Adverse events (AEs) during neoadjuvant treatment, surgery, chemotherapy, and maintenance therapy, grading based on NCI-CTCAE v5.0 (National Cancer Institute-Common Terminology Criteria for Adverse Events Version 5.0). AEs are generally graded from 1 to 4, with higher grades indicating more worse conditions.
Tolerability evaluation | From the start of neoadjuvant therapy to the end of maintenance therapy, assessed up to 30 months.
  The proportion of dose interruptions, dose reductions, and dose discontinuations due to drug-related toxicities during the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Beihua Kong, Principal Investigator — Qilu Hospital of Shandong University; Kun Song, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China